CLINICAL TRIAL: NCT05873166
Title: Stabilometry After Pressure Release of the Flexor Digitorum Brevis Muscle Versus a Non-emission Laser: Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Head of Podiatry, Principal Investigator, and Physiotherapist., Mayuben Private Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1912202200923-A
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Flatfoot
Keywords: Foot; stabilometry; trigger point
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral pressure release in Flexor Brevis Digitorum in subjects with latent trigger point (Experimental): Bilateral pressure release in Flexor Brevis Digitorum in subjects with latent trigger point
  Interventions: Other: Bilateral pressure release in Flexor Brevis Digitorum in subjects with latent trigger point
- Bilateral non emission Laser in latent trigger points of the Flexor digitorum Brevis Muscle (Sham Comparator)
  Interventions: Other: Bilateral non emission Laser in latent trigger points of the Flexor digitorum Brevis Muscle

INTERVENTIONS:
Other: Bilateral pressure release in Flexor Brevis Digitorum in subjects with latent trigger point — Bilateral pressure release in Flexor Brevis Digitorum in subjects with latent trigger point
  Arms: Bilateral pressure release in Flexor Brevis Digitorum in subjects with latent trigger point
Other: Bilateral non emission Laser in latent trigger points of the Flexor digitorum Brevis Muscle — Bilateral non emission Laser in latent trigger points of the Flexor digitorum Brevis Muscle
  Arms: Bilateral non emission Laser in latent trigger points of the Flexor digitorum Brevis Muscle

SUMMARY:
Thirty-six subjects randomly distributed between a pressure release intervention group and a control group whose intervention is a non-emission laser. All the subjects will be measured before and after the interventions of each group. The measurements will be made on a pressure platform to record the stabilometry variables.

DETAILED DESCRIPTION:
Thirty-six subjects randomly distributed between a pressure release intervention group and a control group whose intervention is a non-emission laser. All the subjects will be measured before and after the interventions of each group. The measurements will be made on a pressure platform to record the stabilometry variables with eyes closed and open.

ELIGIBILITY:
Inclusion Criteria:

* Must have latent trigger point in Flexor Brevis Digitorum muscles with no other pathologies

Exclusion Criteria:

* Previous lower extremities surgery. History of lower extremities injury with residual symptoms (pain, "giving-away" sensations) within the last year.

Leg-length discrepancy more than 1 cm Balance deficits (determined by oral questionnaire regarding falls)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Stabilometry variables eyes open before pressure release (x) | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X (in millimeters) with open eyes.
Stabilometry variables eyes open before pressure release (y) | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in Y (in millimeters) with open eyes.
Stabilometry variables eyes open before pressure release COP area | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of Pressure (COP) area (in millimeters2) with eyes open.
Stabilometry variables eyes open before pressure release COP a-p | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the anteroposterior(a-p) direction (in millimeters/second).
Stabilometry variables eyes open before pressure release COP lat-lat | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the latero-lateral(lat-lat) direction (in millimeters/second).
Stabilometry variables eyes closed after pressure release (x) | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X (in millimeters) with eyes closed.
Stabilometry variables eyes closed after pressure release (y) | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in Y (in millimeters) with closed eyes.
Stabilometry variables eyes closed after pressure release COP area | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of Pressure (COP) area (in millimeters²) with eyes closed.
Stabilometry variables eyes closed after pressure release COP a-p | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the anteroposterior(a-p) direction (in millimeters/second).
Stabilometry variables eyes closed after pressure release COP lat-lat | Through study completion, an average of 1 week
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the latero-lateral(lat-lat) direction (in millimeters/second).

CONTACTS AND LOCATIONS:
Overall Officials: Eva María Martínez-Jimenez, PhD, Principal Investigator — Mayuben Private Clinic
Locations (1):
- Eva María Martínez-Jimenez, Madrid, Spain